CLINICAL TRIAL: NCT05098938
Title: A Randomized, Multi-Center, Double Blinded, Self-Initiated, Single Treatment Study Comparing Sitavig® (Acyclovir) 50 mg Muco-adhesive Buccal Tablet to Placebo in the Treatment of Herpes Labialis in Immunocompetent Adults
Brief Title: A Study to Compare Sitavig (Acyclovir) Buccal Tablet With a Placebo in the Treatment of Herpes Labialis in Participants Whose Immune System Works Normally
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21755
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — Acyclovir; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acyclovir 50mg buccal/topical tablet treatment group (Experimental)
  Interventions: Drug: Acyclovir 50mg buccal/topical tablet, BAYM008894/UI1614773
- Matching placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir 50mg buccal/topical tablet, BAYM008894/UI1614773 — Oral (upper gum area), 50mg, 1 tablet.
  Arms: Acyclovir 50mg buccal/topical tablet treatment group
Drug: Placebo — Oral (upper gum area), 1 table.
  Arms: Matching placebo group

SUMMARY:
Researchers are looking for a better way to treat people who have recurrent herpes labialis, also known as cold sores. This is a type of viral infection that causes redness and blisters on the mouth and lip and that recurs.

Herpes labialis is caused by a virus called the herpes simplex virus (HSV). The infection is spread when a person comes into direct contact with someone else who has the infection. Once a person becomes infected with HSV, the virus multiplies and spreads, which can cause redness and blistering on the mouth and lip. The blisters crust over and heal. Once healed, the virus is said to go into an "inactive" phase. This means the virus does not cause any symptoms, but still remains in the body. HSV can then become "active" again. This means causing cold sore lesions to reappear. HSV can become active in different ways. Some of these include when a person has a fever, comes into contact with strong sunlight or has a condition that lowers one's immune system It can also happen during a woman's menstrual cycle, also called a period.

In this study, the researchers want to gather additional data on acyclovir 50 mg tablet, an available treatment for herpes labialis. It is a buccal tablet that sticks to the gum inside the mouth and directly treats the infected area to help stop the HSV from multiplying and spreading.

In this study, the researchers want to compare the efficacy of acyclovir 50 mg buccal tablets versus placebo in the treatment of herpes labialis. A placebo is a treatment that looks like the study medicine but does not have any medicine in it. Study participants will include those who have had at least 4 episodes of herpes labialis within the past 12 months prior to joining the study. To compare the study treatments, the researchers will measure the "duration of episode" (DOE) for each participant. DOE is amount of time it takes for symptoms to disappear and for herpes labialis lesions to heal after taking the study treatment. A doctor will look at the participants' symptom scores and facial images to determine the DOE. Assessments will be done over a period of 14 days.

The participants in this study will apply either acyclovir 50mg buccal tablet or the placebo as a tablet to the upper gum 1 time.

There will be a 2 week treatment phase and a 12 month follow up phase. The participants in this study will not be required to visit the study site. Instead, the participants will have virtual meetings with the study doctors from their homes using the internet. During the treatment phase, there will be 2 meetings. Throughout the follow up phase, the doctors will call the participants 4 times. Each participant will be in the study for about 20 months.

During the treatment phase of the study, the participants will:

* take their blood pressure and pulse
* check their mouth health through a questionnaire
* take pictures of their face and herpes labialis symptoms During the whole study the participants will answer questions about how they are feeling, what medications they are taking, and what adverse events they are having.

The doctors will keep track of any adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

DETAILED DESCRIPTION:
Participants will be randomly assigned one of two treatment groups - acyclovir 50 mg buccal tablet or a placebo buccal tablet. Face images as well as symptom scores will be recorded at baseline, treatment initiation and over the next 14 days. Participants will automatically transition to the Follow-up Phase. Participants will be in contact with the sites using weekly virtual check-ins with the e-diary/App with the purpose reporting any adverse events, concomitant medications , or new outbreaks of herpes labialis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years of age or older inclusive;
* History of recurrent HL lesions where:

  * Recurrence is defined as at least 4 episodes in the preceding 12 months;
  * At least half of the episodes should be vesicular in nature;
  * At least half of the episodes should be preceded by prodromal symptoms;
  * Herpes labialis lesions are characterized by their localization on the cutaneous and/or mucosal surfaces of the lips;
* Willing to avoid, during the treatment phase, the use of anti-inflammatory (not including low-dose (81 mg) aspirin), anti-herpetic, antibiotic and antiviral agents as well as steroids or other natural products that would interfere with the immune system response;
* Female participants of childbearing potential must be using a medically acceptable form of birth control during screening [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier], abstinence or in same sex relationship and have a negative pregnancy test at Screening and prior to study drug administration. Female participants of non-childbearing potential must be amenorrheic for at least two years or have undergone surgical sterilization (i.e. tubal ligation/occlusion, hysterectomy and/or bilateral oophorectomy);
* Agreement to abstain from any mechanical disruption of the prodromal area or lesion (i.e. scrubbing, lancing, shaving the area, rubbing with alcohol, application of heat emitting devices used for cold sore treatment, etc.);
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol;
* Ability to understand and follow study-related instructions;
* Be willing and able to participate in all scheduled visits, treatment plan, and trial procedures according to the clinical protocol.

Exclusion Criteria:

* Participants who did not develop herpes prodromal symptoms within 6 months after randomization in the study;
* More than 50% of recurrences that aborted spontaneously (without intervention) in the past 12 months;
* Primary herpes lesion outside the lips (e.g., nose, chin, etc.);
* Abnormal peri-oral skin condition that might affect the normal course of cold sores (e.g., eczema, psoriasis, etc.);
* Oral diseases whose prodromal symptoms may mimic those of herpes labialis, including recurrent oral aphthous disease;
* Allergy to any acyclovir or its containing agents;
* Milk allergy or known history of hypersensitivity to one of the components of Sitavig;
* Self-reported immunocompromised condition, including self-reported Human Immunodeficiency Virus (HIV) positive and previous bone marrow or organ transplant;
* Known medical history of renal disease, that in the judgment of the investigator is severe;
* Females who are planning to become pregnant, are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2020 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Science 37, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States of America (USA) as a decentralized study between 23 Nov 2021 (First participant first visit) and 2 July 2024 (Last participant last visit).
Pre-assignment Details: 2020 participants were randomized into the study, 1009 in the Sitavig arm and 1011 in the Placebo arm.
  1019 participants were run-in failure, 505 in the Sitavig arm and 514 in the Placebo arm, so that 504 participants were included in the Sitavig arm and 497 in the Placebo arm.
Groups:
- Sitavig: Sitavig (acyclovir) 50 mg muco-adhesive buccal tablet (one tablet application on Day 1)
- Placebo: Placebo muco-adhesive buccal tablet (one tablet application on Day 1)
Period: Overall Study
Arm/Group | Sitavig | Placebo
Started | 1009 | 1011
Completed | 372 | 369
Not Completed | 637 | 642
Not completed — Adverse Event | 4 | 3
Not completed — inclusion/exclusion criteria change | 11 | 5
Not completed — lack of compliance | 26 | 19
Not completed — Lost to Follow-up | 37 | 40
Not completed — Lost in treatment period | 17 | 13
Not completed — Met an exclusion criterion | 0 | 3
Not completed — no prodromal symptoms after 6 months | 1 | 0
Not completed — Physician Decision | 25 | 32
Not completed — Run in failure in treatment phase | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Run-in Failure in early study | 505 | 514
Not completed — IMP delivery missed | 1 | 5
Not completed — 6 months visit was missed | 2 | 0
Not completed — fit for use was not completed within window | 3 | 0
Not completed — V2 visit was not completed within window | 0 | 1
Not completed — exclusionary medication use | 1 | 2
Not completed — change in medication | 1 | 0
Not completed — treatment failure | 2 | 1

BASELINE CHARACTERISTICS:
Population: The demographic and baseline characteristics were summarized for the Intent-to-treat population, i.e. all participants who were randomized and provided at least one measure of primary efficacy parameters after the first dose of study intervention i.e., if there was at least one non-missing assessment of participant's face image using a 6-point Likert scale after study intervention initiation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitavig | Placebo | Total
Number analyzed (Participants) | 493 | 483 | 976
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (12.38) | 43.0 (12.19) | 42.9 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 402 | 399 | 801
  Male | 91 | 84 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 37 | 80
  Not Hispanic or Latino | 450 | 445 | 895
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Episode (DOE) Was Measured in Hours (Using the Science 37 Platform), of a Single Treated Herpes Labialis (HL) Lesion
Description: Duration of episode (DOE) is defined as the time from the initiation of treatment (study intervention) to the healing of primary lesions (loss of crust) for participants who experience a vesicular lesion.
  For participants whose primary lesions are not vesicular in nature, duration of episode is the time from study intervention initiation to the return to normal skin as determined by the independent blinded reader of the participant's face images using a 6-point Likert scale or to the cessation of symptoms, whichever comes last.
Time Frame: Up to 14 days
Population: PP population: The Per Protocol (PP) population included all subjects who completed 14-days of evaluations and did not have any major protocol violations.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 330 | 349
Hours | 66.5 [55.4 to 74.7] | 73.6 [65.5 to 85.2]
Statistical Analysis 1: Comparison: Sitavig vs Placebo; Test type: Superiority; p = 0.716, Log Rank

2. Secondary Outcome: Incidence of Aborted Lesions
Description: Incidence of aborted lesions, defined as treated HL lesions that do not progress to the vesicular or crust stage. A lesion that returns to normal skin without forming a vesicle or crust will be counted as an aborted lesion.
Time Frame: Up to 14 days
Population: PP population: The Per Protocol (PP) population included all subjects in ITT who completed 14-days of evaluations and did not have any major protocol violations.
Measure: Number; unit: lesions
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 330 | 349
lesions | 40 | 58
Statistical Analysis 1: Comparison: Sitavig vs Placebo; Test type: Superiority; p = 0.102, Chi-squared

3. Secondary Outcome: Incidence of Recurrence of HL Lesions During the 12-months Follow-up Period
Time Frame: Up to 12 months
Population: Follow-up population: The follow-up population included all participants, who continued into the 12-months Follow-up period and was defined as participants whose lesions were all treated at the end of the treament period (of 14 days) of the study.
Measure: Number; unit: lesions
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 378 | 400
lesions | 117 | 94
Statistical Analysis 1: Comparison: Sitavig vs Placebo; Test type: Superiority; p = 0.712, Chi-squared

4. Secondary Outcome: Time to Recurrence of HL Lesions, Measured in Days From Resolution of the Cold Sore Treated in the Treatment Phase Until Onset of Prodromal Symptoms
Time Frame: Up to 12 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 378 | 400
days | 88.0 [63.0 to 108.0] | 88.0 [65.0 to 106.0]
Statistical Analysis 1: Comparison: Sitavig vs Placebo; Test type: Superiority; p = 0.575, Log Rank

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAE)s
Time Frame: Up to 12 months
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 504 | 497
participants
  Participants with TEAEs | 146 | 149
  Participants with serious TEAEs | 4 | 6
  Participants with treatment related TEAEs | 16 | 10
  Participants with treatment related serious TEAEs | 0 | 0
  Participants with TEAEs leading to study discontinuation | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Have at Least One Recurrence
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Sitavig | Placebo
Number analyzed (Participants) | 378 | 400
percentage of participants | 31.0 | 23.5

ADVERSE EVENTS:
Time Frame: From signing of the consent form until 12 months after end of study intervention, up to 18 months.
Description: Adverse Events were collected on the Safety Population, i.e. all randomized participants who took at least one dose of study intervention.
Arm/Group | Sitavig | Placebo
All-Cause Mortality (participants affected / at risk) | 1/504 | 0/497
Serious Adverse Events (participants affected / at risk) | 5/504 | 7/497
Other Adverse Events (participants affected / at risk) | 143/504 | 146/497
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitavig (N=504) | Placebo (N=497)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Hernia hiatus repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitavig (N=504) | Placebo (N=497)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Aspiration joint (Investigations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 0 (0)
Biopsy muscle (Investigations) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 23 (23) | 27 (28)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dental caries (Gastrointestinal disorders) | 3 (4) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 5 (5) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Gingival discomfort (Gastrointestinal disorders) | 2 (3) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 2 (2)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 2 (2) | 2 (2)
Implant site rash (General disorders) | 1 (1) | 0 (0)
Implant site ulcer (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 9 (9)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Laparoscopic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 2 (2) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
Morton's neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 10 (10)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 3 (3) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Overgrowth bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 6 (6)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinophyma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seasonal affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 9 (9) | 9 (11)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (19) | 20 (21)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (8)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Initial results (Feb 2024) indicated significant data inconsistencies. After quality analysis of the data, it appears that the contract research organization (CRO) did not read the facial images correctly, which are the data source for the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per Master Service Agreement between Bayer and Science 37 dated 08-Apr-2019, Science 37 shall have no rights of publication whatsoever in connection with the Study nor will Science 37 assist any other Party in the preparation of a publication. Publication of results in whole or in part, shall be within the sole and absolute discretion of Bayer, and such shall not be unreasonably withheld.

DOCUMENTS (2):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT05098938/Prot_004.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05098938/SAP_005.pdf